CLINICAL TRIAL: NCT01901822
Title: Root Coverage With Acellular Dermal Matrix Using the Coronally Positioned Tunnel Technique Comparing Two Different Suturing Techniques.
Brief Title: Root Coverage Comparing Suturing Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.0332
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Root Coverage
Keywords: acellular dermal matrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sutured separately (Active Comparator): The soft tissue and the allograft will each be sutured separately using a continuous sling suture.
  Interventions: Procedure: Sutured separately
- Sutured together (Experimental): The soft tissue and the allograft will be sutured together using a continuous sling suture.
  Interventions: Procedure: Sutured together

INTERVENTIONS:
Procedure: Sutured together — The soft tissue and the allograft will be sutured together using a continuous sling suture.
  Arms: Sutured together
Procedure: Sutured separately — The soft tissue and the allograft will be sutured separately using a continuous sling suture.
  Arms: Sutured separately

SUMMARY:
The hypothesis of this study is that coronally positioned tunnel with acellular dermal matrix using a continuous sling suture to secure both the graft and the flap will result in better percent root coverage compared to the continuous sling suturing technique to secure the graft and the flap separately.

DETAILED DESCRIPTION:
Thirty patients will be selected by meeting the following criteria:

Inclusion Criteria:

A. At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985). B. The mucogingival defect must be on a non-molar tooth. C. Patients must be between ≥ 18 years of age.

Exclusion Criteria:

A. Patients with debilitating systemic or diseases that significantly affect the periodontium.

B. Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).

C. Patients requiring antibiotic prophylaxis. D. Root surface restorations at the site of recession. E. No detectable cemento-enamel junction. F. Patients who fail to maintain oral hygiene levels of at least 80% plaque free surfaces.

G. Patients who are pregnant or lactating. H. Patients who use tobacco products (smoking or smokeless tobacco). I. Patients with alcohol abuse problems. J. Patients undergoing long-term steroid therapy. K. History of previous root coverage procedures, graft or guided tissue regeneration, on the test teeth.

L. Patients who fail to complete the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985).
* The mucogingival defect must be on a non-molar tooth.
* Patients must be between ≥ 18 years of age.

Exclusion Criteria:

* Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).
* Patients requiring antibiotic prophylaxis.
* Root surface restorations at the site of recession.
* No detectable cemento-enamel junction.
* Patients who fail to maintain oral hygiene levels of at least 80% plaque free surfaces.
* Patients who are pregnant or lactating.
* Patients who use tobacco products (smoking or smokeless tobacco).
* Patients with alcohol abuse problems.
* Patients undergoing long-term steroid therapy.
* History of previous root coverage procedures, graft or guided tissue regeneration, on the test teeth.
* Patients who fail to complete the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percent root coverage | 6 months
  The amount of root coverage will be measured and converted to a percent.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic University of Louisville, Louisville, Kentucky, United States